CLINICAL TRIAL: NCT03244566
Title: The Utility of Positron Emission Tomography (PET) in Predicting Cervical Lymphatic Metastasis for Mid-lower Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: PET in Guiding Cervical Lymphadenectomy (ECTOP-2003)
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Chief,department of thoracic surgery, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: PETCLM
Record Dates: First submitted 2017-08-06; First posted 2017-08-09 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Cancer
Keywords: positron emission tomography; cervical lymphatic metastasis
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: positron emission tomography — patients who had esophagectomy with 3-field lymphadenectomy underwent examination of positron emission tomography prior to surgery within 2 weeks.

SUMMARY:
Esophageal cancer is the eighth most common cancer around the world, with more than 450000 new cases per year. Esophagectomy with radical lymphadenectomy (2-field lymphadenectomy) is the mainstay of treatment in many countries for patients with esophageal cancer. To improve the survival, 3-field lymphadenectomy combined with cervical lymphadenectomy was started in 1980s. More potential positive lymph nodes were found during more extended lymphadenectomy, offering more accurate TNM staging, affecting consequent treatment. However，3-field-lymphadenectomy was associated with increased surgical morbidity and mortality. Positron emission tomography (PET) is used for detecting distant metastases and lymphatic involvement. The aim of the study is to evaluate the role of PET in predicting cervical lymph metastases of patients with thoracic esophageal squamous cell carcinoma, and to determine if investigators can use PET to guide future cervical lymphadenectomy. (Eastern Cooperative Thoracic Oncology Projects 2003, ECTOP-2003)

DETAILED DESCRIPTION:
From June, 2018, a total of 110 patients with thoracic esophageal carcinoma will be recruited in 4 hospital in China. Participants with resectable esophageal cancer will have PET/CT scan before three-field lymphadenectomy. Lymph nodes will be recored according to the anatomy site. Lymph nodes metastasis diagnosed by PET/CT and by postoperation pathological examination will be compared to evaluate the role of PET/CT in guiding the extent of lymphadenecomy and surgical approach.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven esophageal cancer
2. Resectable cT1-T3/N0-N1 thoracic，operable esophageal lesion. Staging investigations including esophagogastroscopy, chest and abdominal CT scan, and barium swallow
3. Karnofsky performance status greater than or equal to 80%
4. Acceptable pulmonary and cardiac function.
5. Acceptable hepatic, renal and bone marrow function

Exclusion Criteria:

1. Low performance status(Karnofsky score <80%)
2. Past history of malignancy
3. Unresectable advanced disease(T4 or M1a,M1b)
4. Patients with any other serious underlying medical condition that would impair the ability of the patient to receive or comply with protocol treatment
5. Medically unfit for surgical resection
6. Pulmonary reserve inadequate to undergo thoracotomy and extensive mediastinal lymphadenectomy.
7. A significant history of unstable cardiovascular disease that in the opinion of the treating physician should preclude the patient from protocol treatment.
8. Uncontrolled diabetes mellitus or uncontrolled infection, including HIV or interstitial pneumonia or interstitial fibrosis.
9. Significant psychiatric illness that would interfere with patient compliance
10. Severe hepatic cirrhosis or with serious renal disease unacceptable for surgery
11. Salvage surgery after definitive chemoradiotherapy
12. Patients have neoadjuvant chemoradiotherapy
13. Above the age of 80 years
14. Unreliable for follow up

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients had resectable thoracic esophageal squamous cell carcinoma.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
cervical lymph node metastasis | Decembear 2018
  postoperative pathological examination

SECONDARY OUTCOMES:
mediastinal and abdonimal lymph nodes metastasis | Novermber 2018
  postoperative pathological examination
postoperative complications | March 2019
  surgical morbidity and mortality
diseases-free survival | November 2021
  from the time of surgery to the time of first recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, MD, Principal Investigator — Fudan University
Locations (4):
- China (4):
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Fujian Medical University Cancer Hospital, Fuzhou, Fujian
  - Jiangdu people's hospital of Yangzhou, Yangzhou, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai